CLINICAL TRIAL: NCT07077798
Title: Adjuvant Sintilimab Plus Lenvatinib for HCC Characterized With VETC Following Liver Resection: A Multicenter Prospective Study
Brief Title: Adjuvant Sintilimab Plus Lenvatinib for HCC Characterized With VETC Following Liver Resection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wan-Guang Zhang (Other)
Responsible Party: Sponsor-Investigator, Wan-Guang Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHALLENGE-02
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: HCC; VETC; Recurrence; PD-1; Lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — sintilimab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant group (Experimental): Patients in the adjuvant therapy group received PD-1 monoclonal antibody with Lenvatinb adjuvant therapy after liver resection.
  Interventions: Drug: Sintilimab; Drug: Lenvatinib
- Control group (No Intervention): The control group patients did not receive any intervention and were actively monitored after surgery.

INTERVENTIONS:
Drug: Sintilimab — Patient receives first adjuvant sintilimab 2-4 weeks postoperatively, 200 mg IV, every 21 days for a total of 8 cycles
  Arms: Adjuvant group
Drug: Lenvatinib — lenvatinib is initiated orally(12 mg for body weight >= 60kg, 8 mg for body weight < 60kg daily), 2-4 weeks postoperatively for 6 months.
  Arms: Adjuvant group

SUMMARY:
Vessels that encapsulate tumor clusters (VETC) are a novel invasive metastatic factor in hepatocellular carcinoma (HCC), operating independently of the epithelial-mesenchyme transition (EMT). The presence of VETC is associated with a higher rate of postoperative recurrence in HCC patients, indicating a more aggressive biological behavior.Improving the prognosis for VETC-positive patients is a critical issue in clinical oncology.

DETAILED DESCRIPTION:
Previous studies have established that VETC is a novel mode of metastasis, independent of EMT, and may be associated with immune suppression and poor prognosis. Numerous retrospective studies have found that patients with VETC positivity have higher rates of postoperative recurrence and distant metastasis. How to improve the surgical prognosis for VETC-positive patients remains to be explored. Currently, there are no published studies on how to improve the prognosis for this group of individuals. One of our unpublished retrospective studies found that treatment with PD-1 monoclonal antibodies does not effectively improve the prognosis for VETC-positive patients. However, the combination of PD-1 monoclonal antibodies with lenvatinib can effectively reduce postoperative recurrence and improve prognosis in VETC-positive patients. Therefore, we have designed this multicenter, randomized controlled trial to explore the efficacy and safety of lenvatinib in combination with sintilimab in VETC-positive HCC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years;

  * No previous local or systemic treatment for hepatocellular carcinoma;

    * Child-Pugh liver function score ≤ 7; ④ECOG PS 0-1; ⑤BCLC stage 0-C, underwent R0 resection and confirmed by pathology as hepatocellular carcinoma; ⑥No major systemic diseases, immunodeficiency diseases, etc.; ⑦CD34 immunohistochemical staining confirms the presence of VETC in the intratumoral vascular pattern (part or all of the field of view)

Exclusion Criteria:

* Pregnant or breastfeeding women;

  * Recurrent HCC, distant metastasis or other systemic tumors;

    * Vascular invasion involving the mesenteric vein, main portal vein, hepatic vein or inferior vena cava;

      * History of gastrointestinal bleeding within the past 4 weeks;

        * Active infection; ⑥Other significant clinical and laboratory abnormalities that affect safety evaluation; ⑦Inability to follow the study protocol, receive treatment or follow-up as scheduled

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From date of include in this research until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 60 months
  DFS defined as time to recurrence or death after surgery.

SECONDARY OUTCOMES:
Overall survival | From date of include in this research until the date of death from any cause, whichever came first, assessed up to 60 months
  OS defined as time to death from any cause after surgery.
Adverse events | Baseline up to 60 months
  The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) as assessed by CTCAE v5.0

IPD SHARING:
Plan to Share IPD: Yes